CLINICAL TRIAL: NCT07144982
Title: Impact of a Brief Perioperative Counselling Session on Parental Awareness of Passive Smoking in Paediatric Ambulatory Surgery: a Single-centre Observational Study
Brief Title: Perioperative Counselling and Parental Awareness of Second-hand Smoke
Status: Completed | Type: Observational
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Michele Carella, MD PhD ESRA-DRA, University of Liege
Other Study IDs: B7072024000085
Record Dates: First submitted 2025-08-14; First posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Secondhand Smoke Exposure
Keywords: Tobacco Smoke Pollution; Child; Secondhand Smoking; Patient Education; Perioperative Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Provide additional information about the group or cohort, including a description of any interventio: Eligible participants were adult parents who declared current tobacco use and were present at their child's ambulatory surgical visit. Exclusions included parents absent on the day of surgery, procedures postponed, or explicit refusal to participate.
  Interventions: Behavioral: Counselling session

INTERVENTIONS:
Behavioral: Counselling session — Each enrolled parent received a single, standardized counselling session (~15 minutes) delivered in the ambulatory unit by a certified tobacco counsellor. The session followed a fixed script and covered: (1) types of tobacco smoke exposure (primary, secondary and tertiary), (2) health consequences for children with emphasis on perioperative respiratory and anaesthetic risks, (3) practical measures to reduce household exposure (smoke-free home/car rules, behavioural strategies), and (4) brief advice on initial cessation steps and referral options. Structured handouts and signposting to support services were offered when appropriate.

SUMMARY:
In a single-centre observational before-after study (n=31 parental smokers), a standardized ~15-minute tobacco-counselling intervention delivered during the paediatric ambulatory pathway significantly increased parental awareness of secondhand-smoke harms (median total score 34→46; p=0.0026). Item-level gains were greatest for perceived anaesthetic risk and misconceptions about tertiary/indirect exposure. Session acceptability was high, but self-reported behavioural change at 30 days was limited. The perioperative consultation is a feasible "teachable moment"; integration with visual aids, objective exposure measures, structured cessation referral and longitudinal follow-up should be considered to translate awareness into sustained exposure reduction.

ELIGIBILITY:
Inclusion Criteria:

* adult parents who declared current tobacco use and were present at their child's ambulatory surgical visit

Exclusion Criteria:

* parents absent on the day of surgery
* procedures postponed
* explicit refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible participants were adult parents who declared current tobacco use and were present at their child's ambulatory surgical visit. Exclusions included parents absent on the day of surgery, procedures postponed, or explicit refusal to participate.
Sampling Method: Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2024-11-07 (Actual); Primary Completion 2025-03-27 (Actual); Study Completion 2025-03-27 (Actual)

PRIMARY OUTCOMES:
60-points score parental awareness | 4 hours
  The primary outcome was change in parental awareness measured by a six-item questionnaire (each item scored 0-10; total range 0-60) administered at baseline (arrival), immediately after counselling, and at 30 days by telephone.

SECONDARY OUTCOMES:
Smoking changes | 30 days
  Self-reported changes in smoking behaviour at 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- Michele Carella, Liège, Belgium

IPD SHARING:
Plan to Share IPD: No